CLINICAL TRIAL: NCT02610075
Title: A Phase Ib Study to Determine the Maximum Tolerated Dose (MTD) of AZD1775 Monotherapy in Patients With Locally Advanced or Metastatic Solid Tumours.
Brief Title: Phase Ib Study to Determine MTD of AZD1775 Monotherapy in Patients With Locally Advanced or Metastatic Solid Tumours.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6015C00003; REFMAL 398 (Other: Sarah Cannon Development Innovations)
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Locally Advanced Solid Tumours; Metastatic Solid Tumours; Ovarian Cancer
Keywords: AZD1775; Metastatic solid tumors; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1775 (Experimental): This is a single-arm study in which all patients will receive AZD1775 orally. Patients will continue to receive treatment with AZD1775 until disease progression, intolerable toxicity, or discontinuation criteria are met.
  Interventions: Drug: AZD1775

INTERVENTIONS:
Drug: AZD1775 — All patients will receive intervention with AZD1775 orally. Patients will continue to receive treatment with AZD1775 until disease progression, intolerable toxicity, or discontinuation criteria are met.

SUMMARY:
This Phase Ib study will identify the Maximum Tolerated Dose (MTD) of AZD1775 monotherapy when administered orally once daily (QD) or two times per day (BID) on Days 1 to 5 followed by 9 days of rest in 14-day cycles, or QD on a 5/2 dosing schedule (5 days on, followed by 2 days rest) in 21-day cycles in patients with locally advanced or metastatic solid tumours. Alternative treatment schedules may be explored if preliminary data suggest these would be more appropriate.

The effect of food on single dose PK of AZD1775 will be assessed in 12 patients. In this sub-study, patients will receive a single oral dose of AZD1775 with 240 mL of water, once in the fasted state and once following a high-fat meal.

DETAILED DESCRIPTION:
This study will attempt to determine the Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of AZD1775 monotherapy when administered orally once daily (QD) or two times per day (BID) on Days 1 to 5 followed by 9 days of rest in 14-day cycles, or QD on a 5/2 dosing schedule (5 days on, followed by 2 days rest) in 21-day cycles in patients with locally advanced or metastatic solid tumours. Both the QD 5/9 and 5/2 dosing schedules will run in parallel. An evaluation will be made after the second QD cohort has been completed to determine whether to proceed with one or both dosing schedules.

The AZD1775 MTD will be determined through dose-escalation using a 3+3 cohort design. If less than one-third of evaluable patients in a given cohort (0 of 3 patients or 1 of 6 patients) experiences a Dose-Limiting Toxicity (DLT); escalation may proceed to the next higher dose level. If one of the first 3 patients enrolled in a given cohort experiences a DLT, 3 additional patents will be enrolled in that cohort. If a DLT is observed in one-third or more of patients, the dose at which this occurs will be considered not tolerated and the MTD will have been exceeded. The highest dose level(s) at which less than one-third of patients (0 of 3 patients or 1 of 6 patients) experiences a DLT will be declared the MTD. Up to 6 patients will be enrolled in each cohort. Dose escalation will continue until identification of the MTD or Sponsor termination of the study.

A maximum of 10 dose escalations are anticipated in the determination of MTD. Approximately 6 subjects may be added to replace non-evaluable patients. Therefore, a total of 66 patients are expected to be treated.

Dose-limiting toxicities will be evaluated during Cycles 1 and 2 of treatment. If appropriate the DLT observation period can be expanded by up to 2 weeks in case of treatment delay due to study drug-related adverse events. Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. Patients must complete Cycle 1 and Cycle 2 safety evaluations which will conclude on Cycle 3 Day 1, and must receive at least 80% of the planned dose to be considered evaluable. Patients receiving less than 80% of Cycle 1 and Cycle 2 dose (28 days) will be replaced unless they experienced a confirmed DLT.

The patient population used to determine the MTD will consist of patients who have met the minimum safety evaluation requirements of the study, and/or who have experienced a DLT in Cycle 1 or Cycle 2. Minimum safety requirements will be met if during Cycle 1 and Cycle 2 of treatment the patient receives a minimum of 80% of treatment doses of AZD1775, completes the safety evaluations, and is observed for at least 28 days. Patients who do not meet these minimum safety evaluation and treatment requirements and whom do not experience a DLT will be replaced.

Patients will be allowed to continue treatment with AZD1775 until evidence of disease progression, unacceptable toxicity, or other discontinuation criterion has occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Prior palliative radiation completed ≥ 7 days prior to the start of AZD1775 and recovered from any acute adverse effects.
2. ECOG PS score 0 or 1.
3. Baseline laboratory values:

   * ANC ≥1500/μL
   * Hemoglobin (HgB) ≥9 g/dL
   * Platelets ≥100,000/μL
   * ALT and AST ≤3 x ULN or ≤5 x ULN if known hepatic metastases.
   * Serum bilirubin WNL or ≤1.5 x ULN in patients with liver metastases; or total bilirubin ≤3.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's Syndrome.
   * Serum creatinine ≤1.5 x ULN, or measured creatinine clearance ≥45 mL/min.
4. Females who are not of child-bearing potential and fertile females of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 3 days prior to, and on the day of starting study treatment.
5. Males willing to use at least one medically acceptable form of contraception for duration of study and for 3 months after treatment stops.
6. Predicted life expectancy ≥12 wks.
7. Age ≥18
8. Histologically or cytologically documented locally advanced or metastatic solid tumour, excluding lymphoma, for which standard therapy does not exist or has proven ineffective or intolerable.
9. Measurable or non-measurable disease according to RECIST v1.1.

Exclusion Criteria:

1. Use of a treatment drug 21 days or 5 half-lives (whichever is shorter) prior to AZD1775. For drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the prior treatment and administration of AZD1775 treatment is required.
2. Use of an investigational drug during the past 30 days or 5 half-lives (whichever is longer) prior to first dose of study treatment.
3. Major surgical procedures ≤28 days of beginning study treatment, or minor surgical procedures ≤7 days.
4. Grade >1 toxicity from prior therapy (except alopecia or anorexia).
5. Inability to swallow oral medications.
6. Palliative radiation therapy completed ≤7 days prior to start of study drug.
7. Known malignant CNS disease other than neurologically stable, treated brain metastases.
8. Rx or non-Rx drugs or products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to dosing and withheld until 2 weeks after the last dose of study drug.
9. Patients should stop using herbal medications 7 days prior to first dose of study treatment.
10. Any of the following cardiac diseases currently or within the last 6 months as defined by New York Heart Association (NYHA) ≥ Class 2.

    * Unstable angina pectoris
    * Congestive heart failure
    * Acute myocardial infarction
    * Conduction abnormality not controlled with pacemaker or medication
    * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
11. History of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected.

11. Mean resting QTc interval >470 msec (as calculated per institutional standards) at study entry obtained from 3 ECGs within 5 minutes or congenital long QT syndrome.

12. Pregnant or lactating. 13. Serious active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment.

14. Presence of other active invasive cancers. 15. Psychological, familial, sociological, or geographical conditions that do not permit compliance with protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicities (DLTs) associated with AZD1775 monotherapy administered once daily (QD) in 14 day cycles (5 days on, followed by 9 days rest) in patients with locally advanced or metastatic solid tumours. | Dose-limiting toxicities will be evaluated during the first 2 cycles (28 days) of AZD1775 monotherapy treatment.
  The MTD will be determined through dose-escalation using a 3+3 cohort design. If less than one-third of evaluable patients in a given cohort (0 of 3 patients or 1 of 6 patients) experiences a DLT; escalation may proceed to the next higher dose level. If one of the first 3 patients enrolled in a given cohort experiences a dose-limiting toxicity (DLT), at least 3 additional patents will be enrolled in that cohort. If a DLT is observed in one-third or more of patients, the dose at which this occurs will be considered not tolerated and the MTD will have been exceeded. The highest dose level(s) at which less than one-third of patients (0 of 3 patients or 1 of 6 patients) experiences a DLT will be declared the MTD.
The incidence of dose-limiting toxicities (DLTs) associated with AZD1775 monotherapy administered once daily (QD) in 21-day cycles (5 days on, followed by 2 days rest) in patients with locally advanced or metastatic solid tumours. | Dose-limiting toxicities will be evaluated during the first cycle (21 days) of AZD1775 monotherapy treatment.
  The MTD will be determined through dose-escalation using a 3+3 cohort design. If less than one-third of evaluable patients in a given cohort (0 of 3 patients or 1 of 6 patients) experiences a DLT; escalation may proceed to the next higher dose level. If one of the first 3 patients enrolled in a given cohort experiences a dose-limiting toxicity (DLT), at least 3 additional patents will be enrolled in that cohort. If a DLT is observed in one-third or more of patients, the dose at which this occurs will be considered not tolerated and the MTD will have been exceeded. The highest dose level(s) at which less than one-third of patients (0 of 3 patients or 1 of 6 patients) experiences a DLT will be declared the MTD.
The incidence of dose-limiting toxicities (DLTs) associated with AZD1775 monotherapy administered twice daily (BID) in 14-day cycles (5 days on, followed by 9 days rest) in patients with locally advanced or metastatic solid tumours. | Dose-limiting toxicities will be evaluated during the first 2 cycles (28 days) of AZD1775 monotherapy treatment.
  The MTD will be determined through dose-escalation using a 3+3 cohort design. If less than one-third of evaluable patients in a given cohort (0 of 3 patients or 1 of 6 patients) experiences a DLT; escalation may proceed to the next higher dose level. If one of the first 3 patients enrolled in a given cohort experiences a dose-limiting toxicity (DLT), at least 3 additional patents will be enrolled in that cohort. If a DLT is observed in one-third or more of patients, the dose at which this occurs will be considered not tolerated and the MTD will have been exceeded. The highest dose level(s) at which less than one-third of patients (0 of 3 patients or 1 of 6 patients) experiences a DLT will be declared the MTD.

SECONDARY OUTCOMES:
Plasma concentration of AZD1775 in fasted condition | Samples for AZD1775 PK analysis (fasted) will be taken on Cycle 1 Day 1 predose & 2 hr postdose, Cycle 1, Day 5 pre-dose & 1, 2, 4, 6, 8, & 10 hr post-dose. Samples will also be collected on Cycle 5, Day 3, 4, or 5 pre-dose & pre-dose every 3-5 Cycles.
  Blood samples for determination of AZD1775 concentration will be collected during dose escalation and dose expansion.
Plasma concentration of AZD1775 when dosed with a high fat meal. | Samples for AZD1775 PK food effect analysis will be taken 4 hours after dosing on Cycle 2 Day 1. Subjects will fast for 10 hours prior to dose and for 4 hours post-dose except for the high-fat meal 30 minutes post-dose.
  Blood samples for determination of AZD1775 concentration will be collected during dose escalation and dose expansion.
The incidence of treatment-emergent adverse events (TEAEs) in patients with locally advanced or metastatic solid tumours. | 6 months
  Treatment-emergent adverse events will be assessed by physical examinations, ECOG performance status, complete blood count (CBC) with differential and platelets, clinical chemistry and haematology, triplicate 12-lead ECG, changes in vital signs, and patient reported symptoms.
Best objective response (OR) to treatment will be assessed by dose level cohort according to RECIST v1.1 in patients with locally advanced or metastatic solid tumours. | 8 weeks
  RECIST v1.1 criteria will be used to assess response to treatment. Tumour imaging studies will be repeated every 4 cycles (8 weeks) to assess response until objective disease progression as defined by RECIST v1.1 or withdrawal from study.
  Categorisation of objective tumour response assessment will be based on the RECIST v1.1 criteria of response: Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD). Target lesion progression will be calculated in comparison to when the tumour burden was at a minimum. In the absence of progression, tumour response will be calculated in comparison to the baseline tumour measurements obtained before starting treatment.
The incidence of QTc interval abnormalities in patients with locally advanced or metastatic solid tumours. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Falchook, MD, Principal Investigator — Sarah Cannon Research Institute HealthOne, Denver, CO
Locations (3):
- United States (3):
  - Research Site, Scottsdale, Arizona
  - Research Site, Denver, Colorado
  - Research Site, Nashville, Tennessee

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6015C00003&attachmentIdentifier=22632305-198c-4520-98dd-19476d4c1c80&fileName=D6015C00003_CSP_Redacted.pdf&versionIdentifier=